CLINICAL TRIAL: NCT06981975
Title: Long-term Outcomes of Different Stents for Benign Biliary Stricture Secondary to Chronic Pancreatitis: A Comparative Study Based on a Large Prospective Cohort
Brief Title: Long-Term Outcomes of Different Stents for Benign Biliary Strictures Caused by Chronic Pancreatitis
Acronym: SOLID
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: SOLID
Record Dates: First submitted 2025-05-10; First posted 2025-05-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pancreatitis; Benign Biliary Strictures; Stenting Treatment; ERCP; ESWL
Keywords: Benign Biliary Strictures; Biliary Stenting; Chronic Pancreatitis; Plastic Stents; Self-Expandable Metallic Stents
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- single plastic stent: This cohort consists of patients diagnosed with chronic pancreatitis who underwent endoscopic biliary stenting using single plastic stents to treat benign biliary strictures.
  Interventions: Device: single plastic stent
- multiple plastic stents: This cohort consists of patients diagnosed with chronic pancreatitis who underwent endoscopic biliary stenting using multiple plastic stents to treat benign biliary strictures.
  Interventions: Device: Multiple plastic stents
- Fully covered self-expanding metal stent: This cohort consists of patients diagnosed with chronic pancreatitis who underwent endoscopic biliary stenting using ffully covered self-expanding metal stent to treat benign biliary strictures.
  Interventions: Device: Fully covered self-expanding metal stents

INTERVENTIONS:
Device: single plastic stent — Endoscopic biliary stenting was performed using standard techniques. The maximum bile duct diameter and length of stricture were measured after visualization on x-ray films by retrograde cholangiography. If necessary, sphincterotomy or dilation of the stricture was performed before insertion of the stent. Endoscopic stenting comprised the placement of a single plastic stent. Stents were exchanged at regular intervals or when signs of stent dysfunction were present. If imaging evaluation demonstrated spontaneous passage of the stent with resolution of the stricture, ERCP for stent retrieval was no longer necessary.
  Other Names: SPS
  Groups: single plastic stent
Device: Multiple plastic stents — Endoscopic biliary stenting was performed using standard techniques. The maximum bile duct diameter and length of stricture were measured after visualization on x-ray films by retrograde cholangiography. If necessary, sphincterotomy or dilation of the stricture was performed before insertion of the stent. Endoscopic stenting comprised the placement of multiple plastic stents. Stents were exchanged at regular intervals or when signs of stent dysfunction were present. If imaging evaluation demonstrated spontaneous passage of the stent with resolution of the stricture, ERCP for stent retrieval was no longer necessary.
  Other Names: MPSs
  Groups: multiple plastic stents
Device: Fully covered self-expanding metal stents — Endoscopic biliary stenting was performed using standard techniques. The maximum bile duct diameter and length of stricture were measured after visualization on x-ray films by retrograde cholangiography. If necessary, sphincterotomy or dilation of the stricture was performed before insertion of the stent. Endoscopic stenting comprised the placement of fully covered self-expanding metal stents (fcSEMS) . Stents were exchanged at regular intervals or when signs of stent dysfunction were present. If imaging evaluation demonstrated spontaneous passage of the stent with resolution of the stricture, ERCP for stent retrieval was no longer necessary.
  Other Names: fcSEMS
  Groups: Fully covered self-expanding metal stent

SUMMARY:
This observational study aims to observe and compare the long-term effectiveness and safety of different types of stents for benign biliary strictures secondary to chronic pancreatitis.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is a debilitating condition that often results in the development of benign biliary strictures (BBS), which significantly contribute to morbidity. BBS are prevalent among a substantial number of CP patients, causing complications such as cholestasis and jaundice. Endoscopic biliary stenting has traditionally been the primary treatment for BBS, initially employing single plastic stents (SPS), which yielded suboptimal outcomes.

Nowadays, fully covered self-expanding metal stents (fcSEMS) and multiple plastic stents (MPS) are considered the first line therapies for BBS caused by CP. However, advancements in lithotripsy and endoscopic retrograde cholangiopancreatography have led to a marked increase in the successful rate of pancreatic duct decompression. This progress necessitates a reevaluation of the effectiveness of SPS.

The objective of this study is to assess and compare the long-term outcomes of various stenting types in patients with BBS due to CP. It is expected that the study's results will provide valuable insights into the optimal stenting strategies for BBS in CP patients. These insights have the potential to greatly influence clinical practice and guide the development of treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis
* Benign biliary strictures secondary to chronic pancreatitis
* Patients who have undergone endoscopic biliary stenting for the management of BBS between January 2011 and December 2021.
* Complete Treatment Records

Exclusion Criteria:

* Patients diagnosed with pancreatic cancer within two years following the diagnosis of CP.
* Incomplete Records of endoscopic biliary stenting treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent endoscopic biliary stenting for the management of Benign biliary strictures secondary to chronic pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2025-05-24 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Long-term clinical success | 14 year follow up
  Being recurrence-free from the time of initial stent removal or spontaneous stent passage

SECONDARY OUTCOMES:
Early clinical success | 1 year since the initial procedure
  Benign biliary stricture resolution within 1 year since the initial procedure
Number of Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures | 14 year follow up
  Number of Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures during the initial treatment period (excluding ERCP treatment after stricture recurrence)
Total number of stents placed | 14 year follow up
  Total number of stents placed during the initial treatment period (excluding stents placed for stricture recurrence)
Total stenting time | 14 year follow up
  Total stents placement duration of the initial treatment period (from stent placement to stent removal or spontaneous passage)
Technical success | 14 year follow up
  Technical success defined as the ability to deploy the stent(s) in satisfactory position during initial stent placement procedure.
Stricture recurrence | 14 year follow up
  Abnormalities in liver function tests and the need for repeat intervention after a period of stent removal
Procedure- or device-related adverse events | 14 year follow-up
  Device or procedure related serious adverse events from the initial stent placement procedure to the 14 year follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haapamaki C, Kylanpaa L, Udd M, Lindstrom O, Gronroos J, Saarela A, Mustonen H, Halttunen J. Randomized multicenter study of multiple plastic stents vs. covered self-expandable metallic stent in the treatment of biliary stricture in chronic pancreatitis. Endoscopy. 2015 Jul;47(7):605-10. doi: 10.1055/s-0034-1391331. Epub 2015 Jan 15. PMID 25590182
- [Background] Cote GA, Slivka A, Tarnasky P, Mullady DK, Elmunzer BJ, Elta G, Fogel E, Lehman G, McHenry L, Romagnuolo J, Menon S, Siddiqui UD, Watkins J, Lynch S, Denski C, Xu H, Sherman S. Effect of Covered Metallic Stents Compared With Plastic Stents on Benign Biliary Stricture Resolution: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1250-7. doi: 10.1001/jama.2016.2619. PMID 27002446
- [Background] Ramchandani M, Lakhtakia S, Costamagna G, Tringali A, Puspoek A, Tribl B, Dolak W, Deviere J, Arvanitakis M, van der Merwe S, Laleman W, Ponchon T, Lepilliez V, Gabbrielli A, Bernardoni L, Bruno MJ, Poley JW, Arnelo U, Lau J, Roy A, Bourke M, Kaffes A, Neuhaus H, Peetermans J, Rousseau M, Reddy DN. Fully Covered Self-Expanding Metal Stent vs Multiple Plastic Stents to Treat Benign Biliary Strictures Secondary to Chronic Pancreatitis: A Multicenter Randomized Trial. Gastroenterology. 2021 Jul;161(1):185-195. doi: 10.1053/j.gastro.2021.03.015. Epub 2021 Mar 17. PMID 33741314